CLINICAL TRIAL: NCT03197818
Title: A 24-week, Double Blind, Double Dummy, Randomized, Multinational, Multicentre, 2-arm Parallel Group,Active Controlled Clinical Trial of Fixed Combination of Beclometasone Dipropionate Plus Formoterol Fumarate Plus Glycopyrronium Bromide Administered Via pMDI (CHF 5993) Versus the Fixed Combination of Budesonide Plus Formoterol Fumarate (Symbicort® Turbuhaler®) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Active Controlled Trial of CHF5993 Pressurized Metered-dose Inhaler ( pMDI) vs Symbicort®Turbuhaler® in Patients With Chronic Obstructive Pulmonary Disease ( COPD)
Acronym: TRIVERSYTI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-5993AA1-14; China (Other: China: Food and Drug Administration); Taiwan (Other: Taiwan : Food and Drug Administration); South Korea (Other: Ministry of Food and Drugs Safety)
Record Dates: First submitted 2017-01-25; First posted 2017-06-23 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Anticholinergics; Triple Combination
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF 5993 100/6/12.5 µg (Experimental): Fixed combination of extrafine beclometasone dipropionate 100 µg plus formoterol fumarate 6 µg plus glycopyrronium bromide 12.5 µg / metered dose (BDP/FF/GB) (Beclometasone dipropionate / Formoterol Fumarate / glycoppyronium Bromide)
  Interventions: Drug: CHF 5993 100/6/12.5 µg
- Symbicort Turbuhaler 160/4.5 µg (Active Comparator): Fixed combination of 160 µg budesonide + 4.5 µg formoterol fumarate (160µg + 4.5 µg expresses the delivered dose; 200 µg + 6 µg expresses the metered dose) ( BUD/FF) (Budesonide/Formoterol Fumarate)
  Interventions: Drug: 160 µg budesonide + 4.5 µg formoterol fumarate

INTERVENTIONS:
Drug: CHF 5993 100/6/12.5 µg — Fixed combination of extrafine beclometasone dipropionate 100 µg plus formoterol fumarate 6 µg plus glycopyrronium bromide 12.5 µg / metered dose
  Arms: CHF 5993 100/6/12.5 µg
Drug: 160 µg budesonide + 4.5 µg formoterol fumarate — Fixed combination of budesonide 160 µg plus formoterol fumarate 4.5 µg
  Arms: Symbicort Turbuhaler 160/4.5 µg

SUMMARY:
The purpose of this study is to demonstrate the superiority of CHF 5993 pMDI (fixed combination of extrafine beclometasone dipropionate plus formoterol fumarate plus glycopyrronium bromide) over Symbicort® Turbuhaler® in terms of pulmonary function, as well as to assess its safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female adults aged > 40 years with a diagnosis of COPD
* Current smokers or ex-smokers
* A post-bronchodilator FEV1 < 50% of the predicted normal value and a post-bronchodilator FEV1/FVC ratio < 0.7 at least 10-15 minutes after 4 puffs (4 x 100 µg) of salbutamol pMDI
* At least one exacerbation in the 12 months preceding the screening visit

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of asthma, history of allergic rhinitis or atopy
* Patients treated for exacerbations in the 4 weeks prior to screening visit
* Patients treated with non-cardioselective ß-blockers in the month preceding the screening visit
* Patients treated with long-acting antihistamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study or if taken as Pro Re Nata
* Patients requiring long term ( at least 12 hours daily) oxygen therapy for chronic hypoxemia
* Known respiratory disorders other than COPD
* Patients who have clinically significant cardiovascular condition

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in pre-dose FEV1(Forced Expiratory Volume within the first second) at week 24 | Baseline to Week 24
  Change from Baseline in pre-dose FEV1(Forced Expiratory Volume within the first second) at week 24
Change from Baseline in 2-hour post-dose FEV1 at week 24 | Baseline to Week 24
  Change from Baseline in 2-hour post-dose FEV1 at week 24

SECONDARY OUTCOMES:
Change from Baseline in pre-dose morning FEV1 and 2-hour post-dose morning FEV1 at week 24 | Baseline to Week 24
  Change from Baseline in pre-dose morning FEV1 and 2-hour post-dose
Time to First COPD exacerbation | Baseline to week 24
  Time to First COPD exacerbation
Rate of COPD exacerbations | Baseline to week 24
  Rate of COPD exacerbations
Change in COPD Assessment Test (CAT) | At all visits (from baseline to Week 24)
  Change in COPD Assessment Test (CAT)

OTHER OUTCOMES:
Adverse Events and Adverse Drug reactions | Screening up to week 24
  Adverse Events and Adverse Drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (66):
- China (43):
  - Chiesi clinical Trial Site 156031, Beijing, Beijing Municipality
  - Chiesi Clinical Trial Site 156026, Beijing, Beijing Municipality
  - Chiesi clinical Trial Site 156017, Beijing, Beijing Municipality
  - Chiesi Clinical Trial Site 156012, Beijing, Beijing Municipality
  - Chiesi Clinical Trial Site 156045, Chongqing, Chongqing Municipality
  - Chiesi Clinical Trial Site 156002, Fuzhou, Fujian
  - Chiesi clinical Trial Site 156024, Foshan, Guangdong
  - Chiesi Clinical Trial Site 156048, Guangzhou, Guangdong
  - Chiesi Clinical Trial Site 156013, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University site 156001, Guanzhou, Guangdong
  - Chiesi Clinical Trial Site 156008, Zhanjiang, Guangdong
  - Chiesi Clinical Trial site 156003, Nanning, Guangxi
  - Chiesi clinical Trial Site 156020, Haikou, Hainan
  - Chiesi Clinical Trial Site 156044, Shijiangzhuang, Hebei
  - Chiesi Clinical Trial Site 156040, Changsha, Hunan
  - Chiesi Clinical Trial Site 156043, Baotou, Inner Mongolia
  - Chiesi Clinical Trial Site 156015, Baotou, Inner Mongolia
  - Chiesi Clinical Trial Site 156004, Huai'an, Jiangsu
  - Chiesi clinical Trial Site 156033, Jiangyin, Jiangsu
  - Chiesi clinical Trial Site 156022, Nanjing, Jiangsu
  - Chiesi Clinical Trial Site 156049, Suzhou, Jiangsu
  - Chiesi Clinical Trial Site 156047, Jiujiang, Jiangxi
  - Chiesi Clinical Trial Site 156041, Nanchang, Jiangxi
  - Chiesi clinical Trial Site 156028, Nanchang, Jiangxi
  - Chiesi Clinical Trial Site 156042, Pingxiang, Jiangxi
  - Chiesi clinical Trial Site 156023, Changchun, Jilin
  - Chiesi Clinical Trial Site 156036, Changchun, Jilin
  - Chiesi clinical Trial Site 156019, Changchun, Jilin
  - Chiesi Clinical Trial Site 156007, Shenyang, Liaoning
  - Chiesi clinical Trial Site 156025, Yinchuan, Ningxia
  - Chiesi Clinical Trial Site 156014, Shanghai, Shanghai Municipality
  - Chiesi clinical Trial Site 156037, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial Site 156005, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial Site 156006, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial Site 156011, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial Site 156038, Shanghai, Shanghai Municipality
  - Chiesi Clinical Trial Site 156039, Taiyuan, Shanxi
  - Chiesi clinical Trial Site 156035, Chengdu, Sichuan
  - Chiesi Clinical Trial Site 156010, Chengdu, Sichuan
  - Chiesi clinical Trial Site 156032, Chongqing, Sichuan
  - Chiesi clinical Trial Site 156034, Tianjin, Tianjin Municipality
  - Chiesi clinical Trial Site 156018, Hangzhou, Zhejiang
  - Chiesi Clinical Trial Site 156046, Linhai, Zhejiang
- South Korea (14):
  - Chiesi Clinical Trial Site 410003, Chuncheon, Gang'weondo
  - Chiesi Clinical Trial Site 410012, Bucheon-si, Gyeonggido
  - Chiesi Clinical Trial Site 410001, Bucheon-si, Gyeonggido
  - Chiesi Clinical Trial Site 410002, Goyang-si, Gyeonggido
  - Chiesi Clinical Trial Site 410005, Jeonju, Jeonrabugdo
  - Chiesi Clinical Trial Site 410008, Seoul, Seoul Teugbyeolsi
  - Chiesi Clinical Trial Site 410007, Seoul, Seoul Teugbyeolsi
  - Chiesi Clinical Trial Site 410004, Seoul, Seoul Teugbyeolsi
  - Chiesi Clinical Trial Site 410006, Seoul, Seoul Teugbyeolsi
  - Chiesi Clinical Trial Site 410009, Gyeonggi-do, Seoul Teugbyeols
  - Chiesi Clinical Trial Site 410010, Daegu, Ulsan
  - Chiesi Clinical Trial Site 410011, Seoul
  - Chiesi Clinical Trial Site 410013, Seoul
  - Chiesi Clinical Trial Site 410014, Seoul
- Taiwan (9):
  - Chiesi Clinical Trial Site 158001, Keelung, Keelung Municipality
  - Chiesi Clinical Trial Site 158004, Kaohsiung City, Penghu
  - Chiesi Clinical Trial Site 158010, Changhua, Taiwan Province
  - Chiesi Clinical Trial Site 158003, Douliu, Yunlin
  - Chiesi Clinical Trial Site 158010, Changhua
  - Chiesi Clinical Trial Site 158006, Kaohsiung City
  - Chiesi Clinical Trial Site 158008, Taichung
  - Chiesi Clinical Trial Site 158005, Taipei
  - Chiesi Clinical Trial Site 158011, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zheng J, Baldi S, Zhao L, Li H, Lee KH, Singh D, Papi A, Grapin F, Guasconi A, Georges G. Efficacy and safety of single-inhaler extrafine triple therapy versus inhaled corticosteroid plus long-acting beta2 agonist in eastern Asian patients with COPD: the TRIVERSYTI randomised controlled trial. Respir Res. 2021 Mar 23;22(1):90. doi: 10.1186/s12931-021-01683-2. PMID 33757520